CLINICAL TRIAL: NCT01761552
Title: A Prospective, Randomized Controlled Trial Comparing Traditional Methods of Neuromuscular Block Reversal to Sugammadex for Extubation in the Operating Room in ASA 4 and 4E Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0513-12-HMO
Record Dates: First submitted 2012-12-20; First posted 2013-01-04 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Neuromuscular Blockade
Keywords: in ASA 4 AND ASA 4E patients
MeSH Terms: interventions — Atropine; Neostigmine

ARMS (2):
- Sugammadex (tradename Bridion) (Experimental)
  Interventions: Drug: Sugammadex Reversal
- Traditional reversal or spontaneous recovery: (Active Comparator): Atropine/Neostigmine: Atropine, 0.02 mg/ kg, and Neostigmine,0.05 mg/kg diluted in 100 ml Normal Saline and given over a 10 min drip. Reversal will be given only recommended if spontaneous recovery has occurred up to the reappearance of T2 (shallow blockade) following rocuronium induced blockade.
  Interventions: Drug: Atropine/Neostigmine

INTERVENTIONS:
Drug: Sugammadex Reversal
  Arms: Sugammadex (tradename Bridion)
Drug: Atropine/Neostigmine
  Arms: Traditional reversal or spontaneous recovery:

SUMMARY:
To demonstrate that the use of Sugammadex enables physicians to perform early extubation in the operating room in ASA 4 & 4E patients

Primary endpoint:

• Extubation in the operating room before transfer to the PACU or ICU versus keeping the patient intubated when transferred.

Secondary endpoints:

• Time to extubation - measure the difference in time from application of the surgical dressing until extubation. Atelectasis - comparison of chest x-rays (CXR): prior to surgery, on admission to PACU or ICU and 24 hours after admission to PACU or ICU (This is the routine practice at Hadassa hospital for ASA IV patients.)

ELIGIBILITY:
Inclusion Criteria:

* ASA 4 AND ASA 4E patients
* Patients scheduled to undergo any bowel, urogenital or orthopedic surgery under general anesthesia where use of neuromuscular blocking agents is indicated. -

Exclusion Criteria:

* Patients ASA 1-3 or 5
* Patients who have a medical condition which precludes extubation at the end of surgery (i.e., mesenteric event, severe hypothermia etc.).
* Presence of an advanced directive to withhold or withdraw life sustaining treatment (i.e. DNR).
* Hypersensitivity to the active substances or to any of the excipients of medications used
* Patients with severe renal impairment (including patients requiring dialysis (CrCl < 30mL/min))
* Patients with severe hepatic impairment
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Extubation in the operating room before transfer to the PACU or ICU versus keeping the patient intubated when transferred. | 24 hours

SECONDARY OUTCOMES:
Time to extubation - measure the difference in time from application of the surgical dressing until extubation. | 24 hours
Atelectasis - comparison of chest x-rays (CXR): prior to surgery, on admission to PACU or ICU and 24 hours after admission to PACU or ICU (This is the routine practice at Hadassa hospital for ASA IV patients.) | 24 hours

OTHER OUTCOMES:
The effect of Sugammadex on cortisol levels | 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yoram G Weiss, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel